CLINICAL TRIAL: NCT03498807
Title: A Comparison of Optimal Positive End Expiratory Pressure Determination Guided by Electrical Impedance Tomography and Conventional Protective Ventilation Tool in Acute Respiratory Distress Syndrome Patients
Brief Title: A Comparison of Optimal PEEP Determination Guided by EIT and Conventional Protective Ventilation Tool in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Ju Hsu (Other)
Responsible Party: Sponsor-Investigator, Hui-Ju Hsu, respiratory therapist, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106094-E
Record Dates: First submitted 2018-04-05; First posted 2018-04-17 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: ARDS; Acute Respiratory Distress Syndrome
Keywords: ARDS; Acute Respiratory Distress Syndrome; PEEP; pressure-volume loop; Positive End-Expiratory Pressure; hysteresis
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Moderate to severe ARDS patient on mechanical ventilation from ER or word transfer ICU.(P/F≦200+PEEP≧ 5cmH20)
Who Masked: Participant
Masking Description: During this period, all patients were total sedation using continuous infusion, to prevent any spontaneous breathing .All patients were ventilated using a ventilator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group_Use Ventilator P/V tool (Experimental): Use the Pressure/Volume Loop
  Interventions: Device: Ventiltor P/V Loop
- Study group_Use EIT (Active Comparator): Use the Electrical Impedance Tomography
  Interventions: Device: Electrical Impedance Tomography

INTERVENTIONS:
Device: Ventiltor P/V Loop — determine the Optimal PEEP and keep 48hr on ARDS patients
  Arms: Control group_Use Ventilator P/V tool
Device: Electrical Impedance Tomography — determine Optimal PEEP and keep 48hr on ARDS patients
  Arms: Study group_Use EIT

SUMMARY:
The study of positive end-expiratory pressure(PEEP) in the setting mode has not yet been conclusive. there are several ways to choose the best positive end-expiratory pressure(PEEP) mode for ARDS patients. In this study ,the investigators selected two best positive end-expiratory pressure(PEEP) assessment methods to compare:

First is using the conventional postive ventilator to choose positive end-expiratory pressure(PEEP) and the new non-invasive electrical impedance tomography(EIT) guided method and evaluation the treatment outcome in moderate and severe acute respiratory distress syndrome patients by using pressure-volume curve guided and electrical impedance tomography guided positive end-expiratory pressure setting. In this project, we utilize a newly available non-invasive method- electric impedance tomography (EIT) and Protective Ventilation to determine the optimal PEEP on ARDS patients required invasive mechanical ventilator support at a medical center medical ICU (MICU) and cardiovascular ICU (CVICU)- the Far Eastern memorial hospital, Taiwan.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS)，over the years in the treatment policy has been confirmed that: with low tidal volume to achieve lung protection strategy and high positive end-expiratory pressure (PEEP), both can effectively reduce the mortality rate. And increase PEEP，the alveolar pressure is greater than the atmospheric pressure when exhaled，So that can be effective expansion of the lungs to avoid spitting at the end of the alveolar collapse.

The study of PEEP in the setting mode has not yet been conclusive. Currently in the clinical situation，there are several ways to choose the best PEEP mode for ARDS patients. In this study the investigators selected two best PEEP assessment methods to compare:

First is using the conventional postive ventilator to choose optimal and the new non-invasive electrical impedance tomography guided method and evaluation the treatment outcome in moderate and severe acute respiratory distress syndrome patients by using pressure-volume curve guided and electrical impedance tomography guided positive end-expiratory pressure setting. In this project, the investigators utilize a newly available non-invasive method- electric impedance tomography (EIT) and Protective Ventilation to determine the optimal PEEP on ARDS patients required invasive mechanical ventilator support in ICU at the Far Eastern memorial hospital, Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe ARDS patient on mechanical ventilation from ER or word transfer ICU. (P/F≦ 200 with PEEP ≥ 5cmH20) (PEEP greater than or equal to 5 cm H2O and Berlin criteria for ARDS)

Exclusion Criteria:

* On pacemaker
* Pregnant
* Thoracic or spinal cord trauma
* Pneumothorax
* Hemodynamic instability
* IICP

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Compare the survival rate between two groups | Compare the survival rate between two groups during 91 days in hospitalization
  Calculate the survival rate

SECONDARY OUTCOMES:
Oxygention improve rate in the hospital | Compare the PaO2/FiO2 ratio after fixed Optimal PEEP 48hrs later
  Calculate PaO2/FiO2 ratio improvement rate in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hou T Chang, doctor, Study Director — Far Eastern Memorial Hospital; Ping H Wang, Bachelor, Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Banqiao Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
Still in the research phase.May be consider later

REFERENCES:
- [Result] Xu L, Wang Z, Li T, Li Z, Hu X, Feng Q, Duan D, Gao X. [Comparison of extracorporeal membrane oxygenation and mechanical ventilation for inter-hospital transport of severe acute respiratory distress syndrome patients]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2014 Nov;26(11):789-93. doi: 10.3760/cma.j.issn.2095-4352.2014.11.005. Chinese. PMID 25399892
- [Result] Pintado MC, de Pablo R, Trascasa M, Milicua JM, Rogero S, Daguerre M, Cambronero JA, Arribas I, Sanchez-Garcia M. Individualized PEEP setting in subjects with ARDS: a randomized controlled pilot study. Respir Care. 2013 Sep;58(9):1416-23. doi: 10.4187/respcare.02068. Epub 2013 Jan 29. PMID 23362167
- [Result] Sahetya SK, Brower RG. Lung Recruitment and Titrated PEEP in Moderate to Severe ARDS: Is the Door Closing on the Open Lung? JAMA. 2017 Oct 10;318(14):1327-1329. doi: 10.1001/jama.2017.13695. No abstract available. PMID 28973075